CLINICAL TRIAL: NCT01507337
Title: An Open Label, Single Dose Trial With Two Groups Comparing the Pharmacokinetics of Liraglutide in Young Versus Elderly Healthy Subjects of Both Sexes
Brief Title: Comparison of the Effect of Liraglutide in Young Versus Elderly Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1327
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly (Experimental)
  Interventions: Drug: liraglutide
- Young (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — A single dose of 1 mg administered subcutaneously (under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the exposure of liraglutide in young versus elderly healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs, and blood and urinary laboratory assessments
* Age, young subjects: age 18-45 years (both incl.)
* Age, elderly subjects: age at least 65 years
* Body Mass Index (BMI) 18-30 kg/m^2 (both incl.)
* Blood pressure, young: Diastolic 50-90 mmHg, systolic 90-140 mmHg
* Blood pressure, elderly: Diastolic 50-95 mmHg, systolic 92-160 mmHg

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal, metabolic, endocrine, haematological, neurological, psychiatric disease, or other major disorders that could interfere with the objectives of the trial, as judged by the investigator
* Impaired renal function
* Any clinically significant abnormal ECG (electrocardiogram)
* Active hepatitis B and/or active hepatitis C
* Positive HIV (human immunodeficiency virus) antibodies
* Febrile illness within 5 days prior to first administration of liraglutide
* History of alcoholism or drug abuse during the last 12 months
* Smoking of more than 10 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-04; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Area under the liraglutide plasma concentration time curve (AUC 0-t)

SECONDARY OUTCOMES:
Area under the liraglutide plasma concentration time curve (AUC 0-infinity)
Cmax, maximum liraglutide plasma concentration
tmax, time to reach Cmax
t½, terminal plasma elimination half-life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Result] Damholt B, Golor G, Wierich W, Pedersen P, Ekblom M, Zdravkovic M. An open-label, parallel group study investigating the effects of age and gender on the pharmacokinetics of the once-daily glucagon-like peptide-1 analogue liraglutide. J Clin Pharmacol. 2006 Jun;46(6):635-41. doi: 10.1177/0091270006288215. PMID 16707410
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com